CLINICAL TRIAL: NCT01175395
Title: An Open-Label Study of the Safety and Tolerability of Combining 20089 (Triamcinolone Acetonide Intravitreal Injection) When Used Adjunctively With Lucentis® 0.5 mg Intravitreal Injection in Subjects With Subfoveal Neovascular AMD
Brief Title: 20089 TA+Lucentis Combo Intravitreal Injections for Treatment of Neovascular Age-related Macular Degeneration (AMD)
Acronym: 20089/Combo
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: ICON Bioscience Inc (Industry)
Responsible Party: Principal Investigator, Jennifer I. Lim, Professor of Ophthalmology, Director of Retina Services, Department of Ophthalmology and Visual Sciences, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-1067
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Age-Related Macular Degeneration; Choroidal Neovascularization
Keywords: Choroidal neovascular membranes; CNV; AMD; Age-relate Macular Degeneration; CNVM; subfoveal
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IBI-20089/Lucentis (Experimental): Alternate treatment of either 6.9 mg IBI-20089/Lucentis or 13.8 mg IBI-20089/Lucentis
  Interventions: Drug: IBI-20089/Lucentis

INTERVENTIONS:
Drug: IBI-20089/Lucentis — Combining a single dose of IBI-20089 (6.9 mg or 13.8 mg) intravitreal injection adjunctively with Lucentis 0.5 mg intravitreal injection at baseline and monthly intravitreal Lucentis injection PRN based on clinical and OCT results.
  Other Names: IBI-20089 (Triamcinolone Acetonide)

SUMMARY:
The primary purpose of this study is to assess the safety & tolerability of an investigational drug 20089 TA (6.9 mg or 13.8 mg) when used adjunctively with Lucentis 0.5 mg in subjects with sub-foveal neovascular AMD.

DETAILED DESCRIPTION:
The study is being done to test the safety and effectiveness of an investigational drug 20089 TA that will be used in combination with Lucentis for the treatment of CNVM. In CNVM, tiny abnormal blood vessels grow through the retinal layers in the eye. These vessels are very fragile and can leak or bleed. The severity of the symptoms depends on the size of the CNVM and its proximity to the macula (the center of visual field). Symptoms may be mild such as a blurry or distorted area of vision, or more severe, like a central blind spot. Although Lucentis has been approved by the U.S. Food and Drug Administration (FDA) for the treatment of CNVM, the study drug 20089 TA has not yet been approved, and therefore is considered an investigational drug.

Triamcinolone Acetonide (TA) is a corticosteroid (an anti-inflammatory drug) that is used to treat many eye diseases, such as: macular edema (where inflammation causes thickening of the macula), diabetic eye disease, and age-related macular degeneration. TA has also been shown to be effective in treating neovascular AMD (also known as "wet AMD") where there is an abnormal growth of blood vessels in the macula.

Study drug 20089 is an experimental form of the corticosteroid, Triamcinolone Acetonide(TA). 20089 is a new slow-release formula (longer lasting) for intravitreal (into the eye) delivery of TA. This drug releases the active agent TA over a period of approximately 6 months thereby allowing for the improvement of inflammation and/or complications following neovascular AMD.

Although intravitreal Lucentis has been shown to prevent the loss of vision in most neovascular AMD patients and help gain visual acuity (how well we can see), results can only be assured if monthly injections are given. Since monthly injections are a burden on the patient and caregiver, attempts are being made to reduce the burden by combining available treatment options. We hope that by combining 20089 TA with Lucentis a decrease in retinal inflammation, closure of the leaky vessels with a decrease in the number of monthly injections could be achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects, 55 years of age and older.
2. Diagnosis of active, subfoveal choroidal neovascular membranes (CNVM) due to age related macular degeneration (AMD)
3. Visual acuity from 20/25 to 20/400 in the study eye.

Exclusion Criteria:

1. Subjects who have received corticosteroids via any route in the past 30 days.
2. In the opinion of the investigator, patient is known to be a steroid-responder.
3. Subjects with a history of uncontrolled glaucoma (Primary or Secondary)
4. History of ocular surgery (invasive or non-invasive) in the past 90 days
5. Intravitreal treatment with an anti-VEGF agent e.g. bevacizumab, ranibizumab, or pegaptanib within 30 days of the enrollment (Day 0) examination.
6. Patients requiring systemic steroids (greater than 15 mg daily by mouth) or systemic immunomodulatory agents.
7. Active ocular or periocular infection (i.e., bacterial, viral, parasitic or fungal) in either eye or a history of herpetic ocular infection in either eye.
8. Media opacity in the study eye precluding observation or photography of the fundus.
9. Any other clinically significant medical or psychological condition that, in the opinion of the Investigator, would jeopardize the safety of the patient or affect the validity of the study results.
10. Participation in a clinical trial of an investigational drug or device within 30 days of the screening visit.
11. Known history of allergy to corticosteroids.
12. Pregnant or lactating women

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer I Lim, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- UIC Eye and Ear Infirmary, Chicago, Illinois, United States

REFERENCES:
- [Derived] Lim JI, Niec M, Wong V. One year results of a phase 1 study of the safety and tolerability of combination therapy using sustained release intravitreal triamcinolone acetonide and ranibizumab for subfoveal neovascular AMD. Br J Ophthalmol. 2015 May;99(5):618-23. doi: 10.1136/bjophthalmol-2014-306002. Epub 2014 Nov 6. PMID 25376617
- See also: UIC-Ophthalmology Home Page — http://www.uic.edu/com/eye/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Sept 2010 to January 2012.
Groups:
- IBI-20089/Lucentis: Alternate treatment of either 6.9 mg IBI-20089/Lucentis or 13.8 mg IBI-20089/Lucentis
  IBI-20089/Lucentis : Combining a single dose of IBI-20089 (6.9 mg or 13.8 mg) intravitreal injection adjunctively with Lucentis 0.5 mg intravitreal injection at baseline and monthly intravitreal Lucentis injection PRN based on clinical and OCT results.
Period: Overall Study
Arm/Group | IBI-20089/Lucentis
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IBI-20089/Lucentis
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Safety & Tolerability of 20089 TA (6.9 mg or 13.8 mg) When Used Adjunctively With Lucentis 0.5 mg in Subjects With Sub-foveal Neovascular AMD
Description: The primary objective is to assess the ocular safety of 20089 TA (6.9 mg or 13.8 mg)treatment in combination with Lucentis.
  The ocular safety endpoints to be assessed include the number of participants with ocular Adverse Events such as: evidence of endophthalmitis, uveitis, ocular hemorrhage, retinal tear or detachment to be assessed during ophthalmic examinations. Elevated IOP as measured by an applanation tonometer at every visit.
Time Frame: 360 Days
Measure: Number; unit: Number-participants with adverse events
Arm/Group | IBI-20089/Lucentis
Number analyzed (Participants) | 10
Number-participants with adverse events | 0

2. Secondary Outcome: To Determine the Number of Retreatments With Lucentis in Eyes Initially Treated With 20089 TA and Lucentis
Description: Because of the combination - 20089/Lucentis - treatment, patients may not require monthly Lucentis injections as is the current standard of care practice for AMD.
Time Frame: 30 to 360 days
Measure: Median (Full Range); unit: retreatments
Arm/Group | IBI-20089/Lucentis
Number analyzed (Participants) | 10
retreatments | 2 [0 to 6]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Number of subjects who developed progression of cataract Number of subjects with intraocular pressure (IOP) elevation above 25 mmHg Number of subjects with any severe ocular adverse event Number of subjects with any severe systemic adverse event
Arm/Group | IBI-20089/Lucentis
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBI-20089/Lucentis (N=10)
fracture of sacrum (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IBI-20089/Lucentis (N=10)
ocular hypertension (Eye disorders) | 7 (7)
subconjunctival hemorrhage (Eye disorders) | 5 (6)
cataract surgery (Eye disorders) | 1 (1)
vitreous floaters (Eye disorders) | 1 (1)
temporal pallor of optic nerve (Eye disorders) | 1 (1) — Secondary and due to retinal atrophy.
posterior vitreous detachment (Eye disorders) | 2 (2)
retinal hemorrhage (Eye disorders) | 1 (1)
infective vaginitis (Reproductive system and breast disorders) | 1 (1) — Unrelated to eye condition or treatment.
ptosis of eyelid (Eye disorders) | 1 (1)
food poisoning (Gastrointestinal disorders) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1)
watery eye (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No